CLINICAL TRIAL: NCT04448106
Title: Clinical Study for Subjects With Osteoarthritis of Knees, Hips, and Shoulders Using a Combination of Intravenous Infusions With Intra-articular Injection of Autologous Adipose Tissue-Derived Mesenchymal Stem Cells (AdMSCs)
Brief Title: Autologous Adipose Tissue-Derived Mesenchymal Stem Cells (AdMSCs) for Osteoarthritis
Acronym: AdMSCs
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celltex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTX0020-002
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis Shoulder
Keywords: Autologous Adipose-derived Stem Cells (AdMSCs)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: The Phase 2 study is an open-label, 6 arms, randomized, control group clinical study conducted in multiple clinical facilities.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and evaluators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 2 Arm 1 - OA Knee (Experimental): 50 subjects receive two doses of 2.0-2.86 x 10^6 cells/kg on days 0 and 6 via intravenous infusion.
  On day 3, each subject will receive a single dose of 1.0-2.86 x 10^6 cells/kg via intra-articular injection into the injured joint.
  Interventions: Biological: Celltex- AdMSCs
- Phase 2 Arm 2 OA Knee (Active Comparator): Control group- 50 subjects receive three doses of 2.0-2.86 x 10^6 cells/kg on day 0, 3, and 6 via intravenous infusion
  Interventions: Biological: Celltex- AdMSCs
- Phase 2 Arm 3 - OA Hip (Experimental): 50 subjects receive two doses of 2.0-2.86 x 10^6 cells/kg on days 0 and 6 via intravenous infusion.
  On day 3, each subject will receive a single dose of 1.0-2.86 x 10^6 cells/kg via intra-articular injection into the injured joint.
  Interventions: Biological: Celltex- AdMSCs
- Phase 2 Arm 4 - OA Hip (Active Comparator): Control group- 50 subjects receive three doses of 2.0-2.86 x 10^6 cells/kg on day 0, 3, and 6 via intravenous infusion
  Interventions: Biological: Celltex- AdMSCs
- Phase 2 Arm 5 - OA Shoulder (Experimental): 50 subjects receive two doses of 2.0-2.86 x 10^6 cells/kg on days 0 and 6 via intravenous infusion.
  On day 3, each subject will receive a single dose of 1.0-2.86 x 10^6 cells/kg via intra-articular injection into the injured joint.
  Interventions: Biological: Celltex- AdMSCs
- Phase 2 Arm 6 - OA Shoulder (Active Comparator): Control group- 50 subjects receive three doses of 2.0-2.86 x 10^6 cells/kg on day 0, 3, and 6 via intravenous infusion
  Interventions: Biological: Celltex- AdMSCs

INTERVENTIONS:
Biological: Celltex- AdMSCs — Autologous adipose-derived stem cells Culture expanded mesenchymal stem cells isolated from a patient's own abdominal fat tissue
  Other Names: AdMSCs

SUMMARY:
This is a phase 2 open-label, 6 arms (1 study group and 1 control group for each joint category), randomized control group clinical study with 300 subjects diagnosed with osteoarthritis of knees (n=100), hips (n=100) and shoulders (n=100). The study subjects will be evaluated for disease-associated severity according to symptoms, such as pain, mobility, daily active life, and functions using arthritis society established specific measurement tools related to the joints (KOOS and KSS for OA-knees: HOOS and HHS for OA-hips and ASES and CSS for OA-shoulders).

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Male or female
* Subjects in study group must have banked AdMSCs at Celltex (already passed communicable disease screen tests for HIV, syphilis and Hepatitis B and C during banking stage)
* Must understand and voluntarily sign an Informed Consent for study participation obtained prior to undergoing any study-specific procedures
* Must be diagnosed as OA-knees, OA-hips, or OA-shoulders by radiographic criteria and physical examination.

Exclusion Criteria:

* Participation in another clinical study (with use of another Investigational Medical Product) within 3 months prior to study treatment start
* Unwillingness or inability to comply with study procedures
* Patients with serious basic diseases that affect survival, including blood diseases, cachexia, active bleeding, severe malnutrition, etc.
* Clinically active malignant disease
* Previous thrombotic disorder
* History of known pulmonary embolism or known secondary anti-phospholipid syndrome
* Known or suspected hypersensitivity to any components used to culture the AdMSCs, e.g. BSA and sulfur-containing products (e.g., DMSO)
* Major trauma or surgery within 14 days of study treatment start
* Mental condition rendering the subject (or the subject's legally acceptable representative[s]) unable to understand the nature, scope and possible consequences of the study
* Alcohol, drug, or medication abuse within one year prior to study treatment start
* Any condition that, in the Investigator's opinion, is likely to interfere with evaluation of the AdMSC therapy or satisfactory conduct of the study
* Irreversible severe end-organ failure, such as heart failure/attack, stroke, liver and renal failure due to other disease conditions
* Patients or family history with a hypercoagulable status, such as protein C/protein S deficiency, factor V Leiden, prothrombin gene mutation, dysfibrinogenemia, etc.
* History of long-term use of immunosuppressive agents
* Organ transplants in the previous 6 months
* Pregnant, breastfeeding, or desire to become pregnant or unwilling to practice birth control during participation in the study duration, unless surgically sterilized or postmenopausal during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
the frequency and nature of adverse events occurring during the study based on the annualized rate of all AdMSC-associated adverse events (AEs) in all subjects. | 12 months
  safety
Any organ damage or safety concerns determined by SMAC 20 blood test. | 12 months
  Safety

SECONDARY OUTCOMES:
Change of Knee injury and Osteoarthritis Outcome Score (KOOS, 0 is the worst and 100 is the best) from the baseline for OA-knee patients | 12 months
  efficacy
Change of Knee Society Score (KSS, 0 is the worst and 100 is the best) from the baseline for OA-knee patients | 12 months
  efficacy
Change of Hip disability and Osteoarthritis Outcome Score (HOOS, 0 is the worst and 100 is the best) from the baseline for OA-hip patients | 12 months
  efficacy
Change of Harris Hip Score (HHS, 0 is the worst and 100 is the best) from the baseline for OA-hip patients | 12 months
  efficacy
Change of the American Shoulder and Elbow Surgeons Shoulder Score (ASES, 0 is the worst and 100 is the best) from the baseline for OA-shoulder patients | 12 month
  efficacy
Change of Constant shoulder score (CSS, 0 is the worst and 100 is the best) from the baseline for OA-shoulder patients | 12 months
  efficacy
changes in joint images (X-ray or MRI) from the baseline | 12 months
  efficacy

OTHER OUTCOMES:
Number of patients achieve visual analog scale (VAS) pain improvement above 30%, 50% and 70% from the baseline | 12 months
  efficacy
Number of patient achieve Image (X-ray or MRI) improvement above 30%, 50% and 70% from the baseline | 12 months
  efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Derek W Guillory, MD., Principal Investigator — Root Causes Medicine
Locations (1):
- Stanley C Jones, Houston, Texas, United States